CLINICAL TRIAL: NCT02533102
Title: Evaluation of E7050 Pharmacokinetics After 100 mg Single Oral Doses Under Fed and Fasted Conditions and Characterization of E7050 Pharmacokinetics After 100 mg, 200 mg and 400 mg Single Oral Doses Under Fasted Condition in Healthy Subjects
Brief Title: Pharmacokinetics and Food Effect of Single Oral Dose of E7050 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7050-E044-004
Record Dates: First submitted 2015-08-24; First posted 2015-08-26 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Healthy Subjects
Keywords: Pharmacokinetics; E7050; Healthy Subjects
MeSH Terms: interventions — N-(2-fluoro-4-((2-(4-(4-methylpiperazin-1-yl)piperidin-1-yl)carbonylaminopyridin-4-yl)oxy)phenyl)-N'-(4-fluorophenyl)cyclopropane-1,1-dicarboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part A: E7050 100 mg tablet under fasted conditions (Experimental): Participants will receive a single tablet containing 100 mg E7050 following an overnight fast.
  Interventions: Drug: E7050
- Part A: E7050 100 mg tablet with low-fat breakfast (Experimental): Participants will receive a single tablet containing 100 mg E7050 with a standard low-fat meal.
  Interventions: Drug: E7050
- Part A: E7050 100 mg tablet with high-fat breakfast (Experimental): Participants will receive a single tablet containing 100 mg E7050 with a standard high-fat meal.
  Interventions: Drug: E7050
- Part B: E7050 200 mg tablet under fasted conditions (Experimental): Participants will receive a single dose of 200 mg (two 100 mg tablets) of E7050 under fasted conditions.
  Interventions: Drug: E7050
- Part B: E7050 400 mg tablet under fasted conditions (Experimental): Participants will receive a single dose of 400 mg (four 100 mg tablets) of E7050 under fasted conditions.
  Interventions: Drug: E7050

INTERVENTIONS:
Drug: E7050 — 100 mg tablet administered orally

SUMMARY:
This study is designed to first evaluate the effect of food on E7050's pharmacokinetic parameters following the administration of single 100 mg oral doses of E7050 tablet to each normal healthy participant in the study (Part A), and second to characterize E7050 pharmacokinetics after single doses at 200 mg and 400 mg under fasted conditions (Part B). Part A will be a randomized, single-dose, open-label, three-treatment period crossover study. Part B is a nonrandomized, open-label, two-treatment sequential study design. Twelve participants in Treatment Period 1 will receive a single dose of 200 mg of E7050 under fasted conditions. Following review of safety data of the 200 mg dose level, an additional 12 subjects will then receive a single dose of 400 mg of E7050 in Treatment Period 2.

ELIGIBILITY:
Inclusion criteria:

Subjects must meet all of the following criteria to be included in this study:

1. Normal healthy adult males and females (age 18-45 years).
2. Body Mass Index (BMI) greater than or equal to 18 and less than or equal to 32 at the time of Screening.
3. Pregnancy or lactation. Female patients of childbearing potential must have a negative pregnancy test before inclusion into the study, and must agree to use medically acceptable methods of contraception (eg, abstinence, condom + spermicide, or a double-barrier method [eg, condom + diaphragm with spermicide], or intrauterine device (IUD), or have a vasectomised partner) starting at Screening and throughout the entire study period and for 2 months after the last dose of study drug. Those female patients using hormonal contraceptives must also be using an additional approved method of contraception (as described previously) starting at Cycle 1 Day 1, and continuing throughout the entire study period and for 2 months after the last dose of study drug. Postmenopausal women must have been amenorrheic for at least 12 consecutive months; otherwise a pregnancy test is required. Male patients must agree to use contraceptive methods (eg, abstinence, condom + spermicide or a double-barrier method [eg, condom + partner diaphragm with spermicide]).
4. Non-smokers.
5. Willing and able to comply with all aspects of the protocol.
6. Provide written informed consent.

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from this study:

1. Evidence of clinically significant cardiovascular, hepatic, gastrointestinal, renal, respiratory, endocrine, hematological, neurological, or psychiatric disease or abnormalities or a known history of any gastrointestinal surgery that could impact the pharmacokinetics of study drug.
2. Clinically significant illness within 8 weeks or a clinically significant infection within 4 weeks of dosing.
3. Evidence of organ dysfunction or any clinically significant deviation from normal in their medical history.
4. Evidence of clinically significant deviation from normal in physical examination, vital signs, or clinical laboratory determinations at Screening or Baseline.
5. An interval corrected for heart rate (QTcF) interval greater than 450 msec at Screening or Baseline.
6. Females who are either pregnant or lactating.
7. A known or suspected history of drug or alcohol abuse within 6 months prior to screening, or who have a positive urine drug test or alcohol test at Screening or Baseline.
8. Positive results for Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody (HCV) screen.
9. Diagnosis of acquired immune deficiency syndrome (AIDS), or positive test for human immunodeficiency virus (HIV).
10. Participation in another clinical trial less than 4 weeks prior to dosing or current enrollment in another clinical trial.
11. Receipt of blood products within 4 weeks, or donation of blood within 8 weeks, or donation of plasma within 1 week prior to dosing.
12. Hemoglobin level less than 12.0 g/dL.
13. Known history of any significant drug or food allergy or an ongoing seasonal allergy.
14. Use of prescription drugs within 2 weeks prior to Screening (unless drug has a long t1/2, ie, 5 x t1/2 exceeds 2 weeks).
15. Use of over-the-counter (OTC) medications within a minimum of 2 weeks prior to dosing.
16. Requiring a special diet or taking dietary aids known to modulate drug metabolizing enzymes, or who have consumed foods/beverages or herbal preparations containing Kava root, Ginkgo Biloba Extract (GBE), or St. John's Wort within 4 weeks of Baseline Period 1.
17. Known intolerance to the study drug (or any of the excipients).
18. Any medical or other condition which, in the opinion of the investigator, would preclude participation in a clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
E7050 pharmacokinetic parameter: tmax (time to maximum plasma concentration) | 0 hour to 168 hours
E7050 pharmacokinetic parameter: Cmax (maximum observed plasma concentration) | 0 hour to 168 hours
E7050 pharmacokinetic parameter: t lag (time point immediately prior to the first quantifiable concentration) | 0 hour to 168 hours
E7050 pharmacokinetic parameter: AUC 0-t (area under the plasma concentration-time profile from time 0 to the last measurable concentration) | 0 hour to 168 hours
E7050 pharmacokinetic parameter: AUC 0-inf (area under the plasma concentration-time profile from time 0 to infinity) | 0 hour to 168 hours
E7050 pharmacokinetic parameter: t1/2 (the terminal half-life) | 0 hour to 168 hours

SECONDARY OUTCOMES:
Number of participants as a measure of adverse events (AEs) and serious adverse events (SAEs) | Up to 9 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Zuidlarne, Netherlands